CLINICAL TRIAL: NCT07170605
Title: Implementing a Resilience Program in a Trauma-Informed Preschool Population
Brief Title: The Building Resilience Program: Examining Self-Regulation, Behavior, and Resilience in Under-Resourced Preschoolers With ACEs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Kelle DeBoth Foust, Associate Professor, Cleveland State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2022-23; AOTFIRG23DeBoth (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2025-08-25; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Preschool Age Children; Preschool Education; Adverse Childhood Experience; Mental Health; Resilience; Minority Groups
Keywords: preschool; occupational therapy; ACEs; trauma; resilience; intervention; GAS
MeSH Terms: conditions — Psychological Well-Being; Wounds and Injuries | interventions — Mental Health

STUDY DESIGN:
Intervention Model Description: This study uses a randomized two-group pre-posttest comparison waitlist design. Condition 1 is intervention, and condition 2 is "standard care"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - children receiving the 8-week Building Resilience Program (Active Comparator): Out-of-classroom, small group intervention led by occupational therapists, implementation of the manualized BRP
  Interventions: Behavioral: Mental health, positive coping strategies promoting self-regulation and adaptive skills
- Standard care or school readiness condition (Placebo Comparator): This condition for the waitlist control condition was used to account for positive effects that might have been the result of interactions with an occupational therapist. This was designed specifically NOT to overlap with the constructs of the intervention condition and focused on other, more basic elements of school readiness unrelated to mental health, social emotional learning or trauma.
  Interventions: Other: Standard care/School Readiness Condition

INTERVENTIONS:
Behavioral: Mental health, positive coping strategies promoting self-regulation and adaptive skills — The BRP manual includes eight modules delivered over eight weeks: introduction to resilience, identifying and communicating emotions, emotional regulation, coping strategies for self-regulation (2 parts), breath awareness/meditation, applying positive coping strategies, and review/group session with caregiver. Sessions utilize play as the primary occupation, introducing resiliency concepts through 40-60 minute sessions three times each week to provide repetition and application of concepts with multiple opportunities to review, repeat and apply.
  Each BRP session will be implemented by two occupational therapists, one occupational therapy student, and one YWCA staff member. Group size has been determined to approach therapeutic limits with 8-10 students, requiring this staffing ratio for optimal intervention delivery.
  Other Names: Building Resilience Program
  Arms: Intervention - children receiving the 8-week Building Resilience Program
Other: Standard care/School Readiness Condition — The School Readiness protocol supplements existing preschool curriculum while mitigating positive researcher interaction effects. Sessions start with a song and warm-up, including active listening, sharing and turn-taking while targeting different domains each week: perceptual motor, fine motor (tool use), fine motor (coloring), problem solving, teamwork, coordination and motor planning, problem solving (teams), and gross and fine motor (teams). These skills were selected based on feasibility study observations and designed not to overlap with social-emotional skills embedded in the BRP.
  Arms: Standard care or school readiness condition

SUMMARY:
# Brief Summary

The goal of this clinical trial is to learn if a occupational therapy-led trauma-informed care intervention can improve resilience, self-regulation, coping skills, and emotional health in preschoolers ages 2-4 years from under-resourced neighborhoods with a history of adverse childhood experiences (ACEs) and their caregivers. The main questions it aims to answer are:

* Does the Building Resilience Program (BRP) improve stress management, self-regulation, positive affect, engagement, self-efficacy, coping skills and resilience in preschool children?
* Does the Building Resilience Program (BRP) improve resilience, emotional management, and coping strategies in caregivers?

Researchers will compare the Building Resilience Program group to a school readiness skills comparison group to see if the trauma-informed intervention produces greater improvements in resilience and related outcomes.

Participants will:

* Complete pre- and post-intervention assessments measuring resilience, coping skills, emotional health, occupational engagement, and quality of life
* Attend 40-60 minute group sessions, 3x a week for 8 weeks (children will participate in either the BRP intervention or school readiness comparison group)
* Complete individualized Goal Attainment Scaling to track personal progress (children)
* Attend 2-3 in-person caregiver group sessions during the 8-week intervention period plus pre- and post-intervention meetings (caregivers)
* Complete a program evaluation questionnaire at the end of the study (caregivers)

DETAILED DESCRIPTION:
Background and Rationale Children living in under-resourced, poverty-stricken neighborhoods face significantly higher risks for adverse childhood experiences (ACEs) and trauma. In the East Cleveland, Ohio neighborhoods where this study will be conducted, poverty affects 36.5%- 41.6% of residents respectively, compared to the national average of 11.9%. Among neighborhood children, 52.8% to 54.9% live in poverty, with upwards of 80% being Black minorities. More than half of residents qualify for foodbank benefits and less than half have secure, affordable housing.

ACEs related to poverty and low socioeconomic status include experiencing abuse, neglect, witnessing violence or mental illness, food or housing instability, and incarceration of a parent or caregiver. These experiences can severely impact overall quality of life, mental health, and often lead to developmental delays and long-term effects. When parents themselves were impacted by ACEs, it can lead to intergenerational transmission of negative effects.

The American Academy of Pediatrics has specifically identified the critical need to provide interventions that build resilience and address maladaptive responses due to toxic stress resulting from ACEs. Occupational therapists are particularly well-suited to integrate trauma-informed care (TIC) into service delivery through direct intervention and by embedding strategies within occupational engagement, particularly through play as the primary occupation for young children.

Study Design and Innovation This pilot study builds on a prior feasibility study conducted at the YWCA (Young Women's Christian Association) of Cleveland between April-June 2022. The Building Resilience Program (BRP) manual was originally developed for school-age children with chronic pain and was modified to be age and content appropriate for preschoolers ages 2-4 years with trauma history.

The study employs a randomized two-group pre-posttest comparison waitlist design. Given the maximum enrollment of approximately 40 participants at the YWCA Early Learning Center, the study cannot account for all factors that could introduce bias, but the use of a comparison, non-BRP condition will allow comparison between groups over time and account for potential maturation effects. The comparison group will participate in a basic school readiness skills group that excludes resilience training components to avoid contaminating the intervention protocol while providing similar positive adult interactions that could introduce bias.

Intervention Protocols Included both the Building Resilience Program (BRP) primary intervention and the School Readiness Comparison Protocol. In parallel with participants in the BRP condition, caregivers also participate in 2-3 weekly modules in a separate, caregiver group.

Caregiver Component Based on feasibility study findings showing challenges with weekly caregiver participation, the caregiver requirement has been reduced to 2-3 in-person sessions over 8 weeks, combined with incentives and supports to encourage participation. The BRP manual includes weekly parent activities corresponding with child activities.

Caregiver sessions will be conducted by occupational therapists and occupational therapy students, combining materials for in-person sessions as follows:

1. Pre-intervention meeting: BRP and study description, introduction to resilience, highlights from Inside Out movie, Zones of Regulation overview, Q&A
2. Week 3 session: family resilience, high vs. low resilience, resiliency BINGO activity, Kawa River model, Q&A
3. Week 6 session: adaptive vs. maladaptive behaviors, coping strategies, mindfulness, sensory processing and "sensory solutions," community resources
4. Post-intervention meeting: child and self-advocacy, joint plant activity, program review

Recruitment Strategies

Recruitment lessons learned from the feasibility study have informed enhanced strategies:

1. Extended recruitment period from October-December 2023
2. Multiple meeting options: 18 total meetings (3 evening, lunch, and weekend options offered both in-person and virtually)
3. Comprehensive incentive structure: meals and refreshments at in-person meetings, travel compensation (bus passes), optional childcare, small gift card incentives for families completing consent forms and pre-test packets regardless of meeting attendance
4. Multiple distribution methods: paper packets sent home for families unable to attend meetings, with research team available via telephone or email for questions Previously, for the feasibility study participants were recruited by YWCA staff using classroom apps and paper packets, with caregiver pretest documents completed only when gift card incentives were offered. No caregivers participated in weekly Zoom sessions when no incentives were provided.

Statistical Analysis Plan Child Participants (Aim 1)

Each measure will be treated as a continuous variable with six measurement points (excluding Goal Attainment Scaling documented weekly and analyzed over all 8 weeks of BRP participation). Three primary analyses will be conducted:

1. Intervention Effect for Group A: Repeated Measures MANOVA (multivariate analysis of variance) comparing multiple dependent/outcome variables before and after BRP intervention
2. Intervention Effect for Group B: Repeated Measures MANOVA comparing multiple dependent/outcome variables before and after BRP intervention
3. Combined Intervention Effect: Repeated Measures MANCOVA assessing differences between Groups A and B across all measures following BRP intervention, controlling for school readiness program effects for Group B Goal Attainment Scaling T-scores will be calculated according to best practice protocols, with charts created to visualize changes over time, providing individualized, client-centered program measurement for intervention.

Caregiver Participants (Aim 2) Pre-posttest comparisons will be made using MANCOVA approach for multiple dependent variables, with baseline Social Support Survey Instrument scores included as a covariate to control for social support effects on caregivers' emotion management abilities and adaptive coping skills demonstration.

Implementation Considerations

Anticipated Challenges and Mitigation Strategies

1. Irregular attendance: Intervention provided twice weekly to increase exposure opportunities
2. Recruitment and form completion: Additional incentives available if needed, with flexible meeting scheduling options
3. Unidentified diagnoses in preschool participants: Goal Attainment Scaling will address different performance skills and individualize program goals and activities
4. Language barriers: Adapted materials may be needed for caregivers not speaking English as first language, with YWCA community partner guidance for resolution strategies

Community Partnership The YWCA Early Learning Center serves as the on-site location, providing services to under-resourced families, almost all of whom have experienced homelessness and trauma. The YWCA does not currently provide occupational therapy services, making this collaboration an innovative approach to expanding trauma-informed care access in the community.

This study addresses major obstacles in engaging caregivers from under-resourced families who experience chronic stress due to underemployment, financial instability, unstable housing, unpredictable work schedules, and lack of financial resources including childcare. These caregivers cannot afford to volunteer time and efforts without appropriate supports and incentives.

Theoretical Framework The study is rooted in occupational therapy theory, resilience theory and science, with activities derived from existing literature. The program recognizes play as the primary occupation for preschoolers, introducing resiliency concepts through occupation-based intervention approaches. The trauma-informed care framework guides all intervention delivery, acknowledging the impact of trauma on development and the need for safe, supportive environments that promote healing and growth.

Expected Outcomes and Clinical Implications This pilot study will provide necessary data to understand effects of TIC-based intervention programs implemented by occupational therapists on social, emotional, mental health, coping abilities and life satisfaction in this vulnerable population. Results will inform parameters surrounding program implementation, including successes and challenges encountered, which are important for future effectiveness studies and translation into widespread clinical and community practice.

The study aligns with current funding agency priorities for mental health, resilience and trauma-informed care in pediatric populations, providing pilot data necessary for larger-scale funding applications that would support program implementation across multiple preschools and neighborhoods.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at the YWCA Early Learning Center partner facility, between the ages of 24 months and 66 months at the time of enrollment

Exclusion Criteria:

* limited English-speaking fluency (i.e., required a translator), or parent-reported cognitive delays or medical conditions that would prevent independent participation in the program groups

Ages: 24 Months to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Resilience and Engagement | Measured at baseline, week 8 (end of first intervention and wait-list period), and finally at week 16 (end of second intervention period for the waitlist group and follow-up period for the first intervention group)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Curiosity and Persistence measures (parent proxy report, scores calculated as standardized scores for analysis). Original scoring for all is 1-5 scale (Never, Rarely, Sometimes, Often, Always). Higher scores (always/5) are considered higher and more characteristic of a child with characteristics of being resilient.
Self-Regulation | Measured at baseline, week 8 (end of first intervention and wait-list period), and finally at week 16 (end of second intervention period for the waitlist group and follow-up period for the first intervention group)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Flexibility and Frustration Tolerance measures (parent proxy report, scores calculated as standardized scores for analysis). Original scoring for all is 1-5 scale (Never, Rarely, Sometimes, Often, Always). Higher scores (always/5) are considered higher and more characteristic of a child with characteristics of being resilient.
Emotional Health | Measured at baseline, week 8 (end of first intervention and wait-list period), and finally at week 16 (end of second intervention period for the waitlist group and follow-up period for the first intervention group)
  Measured using NIH Toolbox parent proxy report measures for (1) Positive Affect; (2) Anger; (3) Fear; (4) Sadness. Positive Affect rated on 1-4 scale: (1) Not at all (1) A little bit (2) Somewhat (3) Quite a bit and (4) Very much. Anger rated on 1-3 scale: (1) Never or not true, (2) Sometimes or somewhat true, (3) Often or very true. Fear and Sadness rated on a 0-2 scale, (0) Never or not true, (1) Sometimes or somewhat true, (2) Often or very true. All were converted to standardized scores for analysis according to the NIH Toolbox directions for scoring.
Quality of Life/Life Satisfaction | Measured at baseline, week 8 (end of first intervention and wait-list period), and finally at week 16 (end of second intervention period for the waitlist group and follow-up period for the first intervention group).
  NIH Toolbox measures for General Life Satisfaction parent proxy report measured on a 1-5 scale of (1) Strongly Disagree, (2) Disagree, (3) Neither Agree nor Disagree, (4) Agree, (5) Strongly Agree. All scores converted to standardized scores for analysis according to the NIH Toolbox scoring guide.
Quality of Life (QoL) | Measured at baseline, week 8 (end of first intervention and wait-list period), and finally at week 16 (end of second intervention period for the waitlist group and follow-up period for the first intervention group)
  QoL as measured by parent proxy report on the PedsQL including the following domains: Physical, Emotional, Social, School, and a Composite score. Each of these was rated on a scale of 0-4, (0) Never, (1) Almost Never (2) Sometimes (3) Often (4) Almost Always. Scores were translated into standardized scores for analysis according to PedsQL scoring guidelines.
Individualized Goal Attainment Scaling (GAS) goals | GAS scores recorded at baseline, and then 3x per week for 8 weeks during the intervention condition, and 2x per week during the waitlist control condition, across all GAS categories (behavior, engagement/participation and resilience).
  Goals were created for each individual participant related to: behavior, engagement/participation and resilience. Goal Attainment Scaling (GAS) was used to track progress and attainment throughout the project, recorded by members of the research team. Scoring was consistent with typical GAS ratings: a 5-point scale, ranging from -2 to +2, to assess progress toward a specific goal. The 0 level represents the expected outcome with intervention, while -1 and -2 indicate less-than-expected progress or a return to a baseline, and +1 and +2 show progress that exceeds expectations. These ratings were converted to T-scores for analysis (mean 50, SD 10).

SECONDARY OUTCOMES:
Caregiver - Resilience | Measurements taken and baseline and then post-intervention (either week 8 or 16 depending on group assignment)
  Caregiver resilience measured by Adult Resilience Measure-Revised (ARM-R) total score. Caregivers self-report and rate their agreement with statements on a Likert-type scale, 5-point scale: Responses range from "not at all" to "a lot". For the 17-item version, total scores can range from a minimum of 17 to a maximum of 85. The total score of all items is summed to gain an overall resilience score.
Caregiver Well-Being | Measurement taken at baseline and again post-caregiver intervention at week 8 or week 16, depending on group assignment for their child (caregivers participated in intervention during same 8-week timeframe as their child).
  Caregivers self-reported ratings of well-being on the Caregiver Self-Assessment Questionnaire. 18 questions Yes/No responses. Recorded and then scored according to criteria for standardized score.
Caregiver Perceptions | Caregivers and educators provided consent at baseline, interviews completed after program completed between weeks 16-20, based on scheduling limitations and availability. Interviews schedule for 60 minutes.
  Caregiver and teacher/educator perceptions of the BRP. Caregivers and educators were individually interviewed using an IRB approved, research-designed interview guide, in a 1:1 setting, and scheduled for 60 minutes. Responses were audio recorded as well as transcribed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland State University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
It is a very small data set and there are a select few number of sites that this information could be derived from in the sampling and recruitment community. In addition, I have presented on this topic/study with the community partner named, some of those materials are public, and that information would make it much easier to identify where the data was collected. Because the participants are young children, and have experienced trauma, they are a vulnerable population and therefore producing a data set even with de-identified information, may put them at risk.

REFERENCES:
- [Background] Lynch, B. P., Brokamp, K. M., Scheerer, C. R., Bishop, M., Stauble, L., Hagedorn, B., & Endres, L. (2021). Outcomes of Occupational Therapy in Trauma-Informed Care. Journal of Occupational Therapy, Schools, & Early Intervention, 1-17.
- [Background] Pitt, C., Luger, R., Bullen, A., Phillips, D., & Geiger, M. (2013). Parents as partners: Building collaborations to support the development of school readiness skills in under-resourced communities. South African Journal of Education, 33(4), 1-14.
- [Background] Logan B, Jegatheesan D, Viecelli A, Pascoe E, Hubbard R. Goal attainment scaling as an outcome measure for randomised controlled trials: a scoping review. BMJ Open. 2022 Jul 22;12(7):e063061. doi: 10.1136/bmjopen-2022-063061. PMID 35868829
- [Background] Liu M, Luong L, Lachaud J, Edalati H, Reeves A, Hwang SW. Adverse childhood experiences and related outcomes among adults experiencing homelessness: a systematic review and meta-analysis. Lancet Public Health. 2021 Nov;6(11):e836-e847. doi: 10.1016/S2468-2667(21)00189-4. Epub 2021 Sep 30. PMID 34599894
- [Background] Crouch, E., Jones, J., Strompolis, M., & Merrick, M. (2020). Examining the association between ACEs, childhood poverty and neglect, and physical and mental health: Data from two state samples. Children and Youth Services Review, 116, 105155.
- [Background] Creamer, J., Shrider, E. A., Burns, K., & Chen, F. (2022). Poverty in the United States: 2021. US Census Bureau.
- See also: Study protocols for the Child and Youth Resilience Measure (CYRM) and Adult Resilience Measure (ARM) — https://resilienceresearch.org/

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT07170605/Prot_SAP_000.pdf
  • Informed Consent Form: Parent-Guardian Consent for Child Participation (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT07170605/ICF_001.pdf
  • Informed Consent Form: Caregiver Consent for Self Participation (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT07170605/ICF_002.pdf
  • Informed Consent Form: Child Assent Script (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT07170605/ICF_003.pdf